CLINICAL TRIAL: NCT01106040
Title: A Phase 3, Prospective, Open-Label, Multicenter Comparison Study of Lymphoseek® and Vital Blue Dye as Lymphoid Tissue Targeting Agents in Patients With Known Melanoma or Breast Cancer Who Are Undergoing Lymph Node Mapping
Brief Title: Breast and Melanoma Trial With Lymphoseek to Identify Lymph Nodes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Navidea Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NEO3-09
Record Dates: First submitted 2010-04-14; First posted 2010-04-19 (Estimated); Results first posted 2013-06-03 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Breast Cancer; Melanoma
Keywords: Lymphoseek; Breast Cancer; Melanoma; Experimental
MeSH Terms: conditions — Breast Neoplasms; Melanoma | interventions — technetium-diethylenetriaminepentaacetic acid-mannosyl-dextran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lymphoseek, Lymphatic mapping, Injection (Experimental)
  Interventions: Drug: Lymphoseek

INTERVENTIONS:
Drug: Lymphoseek — The total volume of Lymphoseek injection will be between 0.1 - 1.0 mL.
  Other Names: technetium Tc 99m tilmanocept

SUMMARY:
Data from this pivotal clinical trial will be used to support a marketing application (i.e., NDA) of Navidea's Lymphoseek for use in anatomical delineation of lymphoid tissue (nodes) in the lymphatic pathway draining the primary site of a tumor.

Multicenter, open-label, within-patient comparative study of Lymphoseek and vital blue dye in the detection of excised lymph nodes in patients with known melanoma and breast cancer. All patients will receive a single dose of 50 µg Lymphoseek radiolabeled with 0.5 or 2.0 mCi Tc 99m and vital blue dye.

DETAILED DESCRIPTION:
In patients with primary melanoma and breast cancer, lymph node status is often a strong predictor of outcome and influences the course of treatment a patient may follow after surgery. In an effort to reduce the morbidity and costs of detection of lymph node metastases, surgical oncologists have developed a method by which the sentinel lymph node (SLN; the first node in a draining basin) is identified intraoperatively and removed. This technique, called sentinel node biopsy, has extremely high negative predictive values for melanoma metastases and breast cancer metastases. The two largest trials for melanoma, Morton, et al (2005) and Rossi, et al (2006), reported false negative rates of 6.3% and 14.7%, respectively. Morton, et al (2006), in perhaps the most mature trial reported to date, showed a false negative rate of 3.4%. There is growing evidence that sentinel node biopsy will have a significant impact on the management of melanoma. Sentinel node biopsy also has extremely high negative predictive values for breast cancer metastases; the false-negative rates range from 0% to 9%. There is growing evidence that sentinel node biopsy will have a significant impact on the management of breast cancer. Although the survival and local recurrence studies have yet to be completed, the technique has emerged into common practice.

Intraoperative lymphatic mapping (ILM) with a radiopharmaceutical is a nuclear medicine examination which identifies for the surgeon the first lymph node to receive lymphatic flow from the primary tumor site. This node is removed and analyzed for the presence of malignant cells. By locating the lymph node prior to surgery, a small incision can be used to remove the node and a smaller dissection can be employed. The high negative predictive value of the technique seems to provide an accurate staging procedure and may spare patients who are lymph node negative the morbidity of a complete lymph node dissection. Consequently, staging of melanoma by lymph node mapping and biopsy may be equivalent to regional node dissection without the attendant post surgical morbidity.

An ideal lymph node imaging agent would exhibit rapid clearance from the injection site, rapid uptake and high retention within the first draining lymph node, and low uptake by the remaining lymph nodes. The ideal agent would also have low radiation absorption; high biological safety; convenient, rapid, and stable technetium-99m labeling; and biochemical purity.

Lymphoseek (Technetium Tc 99m diethylenetriaminepentaacetic acid mannosyl dextran, [Tc 99m] DTPA Mannosyl Dextran) is a radiotracer that accumulates in lymphatic tissue by binding to a mannose binding protein that resides on the surface of dendritic cells and macrophages. Lymphoseek is a macromolecule consisting of multiple units of DTPA and mannose, each synthetically attached to a 10 kilodalton dextran backbone. The mannose acts as a substrate for the receptor, and the DTPA serves as a chelating agent for labeling with Tc 99m.

Lymphoseek has a diameter of about 5 nm, which is substantially smaller than current agents used for targeting lymphoid tissue. Lymphoseek's small diameter permits enhanced diffusion into lymph nodes and blood capillaries, resulting in a rapid injection site clearance. Upon entry into the blood, the agent binds to receptors in the liver or is filtered by the kidney and accumulates in the urinary bladder.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has provided written informed consent with HIPAA authorization.
2. The patient is a candidate for surgical intervention, with lymph node mapping being a part of the surgical plan.
3. The patient is at least 18 years of age at the time of consent.
4. The patient has an ECOG performance status of Grade 0 - 2 (see Appendix A).
5. The patient has a clinical negative node status at the time of study entry (i.e. T0-4, N0, M0, see Appendix D and E).
6. If of childbearing potential, the patient has a negative pregnancy test within 72 hours prior to administration of Lymphoseek, has been surgically sterilized, or has been postmenopausal for at least 1 year.

   Melanoma Patients
7. The patient has a diagnosis of primary melanoma. Breast Cancer Patients
8. The patient has a diagnosis of primary breast cancer.
9. Patients with pure ductal carcinoma in situ (DCIS) or non-invasive carcinoma if lymph node biopsy is part of the surgical plan.

Exclusion Criteria:

1. The patient is pregnant or lactating.
2. The patient has clinical or radiological evidence of metastatic cancer including palpably abnormal or enlarged lymph nodes (i.e., all patients should be any T,N0,M0, see Appendix D and E).
3. The patient has a known hypersensitivity to Lymphazurin.
4. The patient has participated in another investigational drug study within 30 days of scheduled surgery.

   Melanoma Patients
5. The patient has a tumor with a Breslow depth less than 0.75mm.
6. Patient has had preoperative chemotherapy, immunotherapy, or radiation therapy.
7. Patient has been diagnosed with a prior invasive melanoma that would occur on the same body region or potentially draining to the same nodal basin or patients with truncal or extremity primary melanoma who has had a prior breast cancer potentially draining to the same axillary nodal basin.
8. Patient has undergone node basin surgery of any type or radiation to the nodal basin(s) potentially draining the primary melanoma.
9. Patient has undergone a wide excision for their primary melanoma (>1 cm in dimension) or complex reconstruction (rotation, free flap, or skin graft of any type).

   Breast Cancer Patients
10. The patient has bilateral primary breast cancers or multiple tumors within their breast.
11. Patient has had prior surgical procedures such as breast implants, reduction mammoplasty, or axillary surgery.
12. Patient is scheduled for bilateral mastectomy unless for cosmetic reasons and the contraindicated breast will not undergo lymph node mapping.
13. Patient has had preoperative radiation therapy to the affected breast or axilla.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2010-06; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon A Blackburn, Study Director — Navidea Biopharmaceuticals
Locations (8):
- United States (8):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - UCSD Moores Cancer Center, La Jolla, California
  - Califonia Pacific Medical Center, San Francisco, California
  - John Wayne Cancer Institute, Santa Monica, California
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - University Hospitals Cleveland, Cleveland, Ohio
  - Breast Care Specialists, Columbus, Ohio
  - The Ohio State University, Columbus, Ohio

REFERENCES:
- [Result] Wallace AM, Han LK, Povoski SP, Deck K, Schneebaum S, Hall NC, Hoh CK, Limmer KK, Krontiras H, Frazier TG, Cox C, Avisar E, Faries M, King DW, Christman L, Vera DR. Comparative evaluation of [(99m)tc]tilmanocept for sentinel lymph node mapping in breast cancer patients: results of two phase 3 trials. Ann Surg Oncol. 2013 Aug;20(8):2590-9. doi: 10.1245/s10434-013-2887-8. Epub 2013 Mar 17. PMID 23504141
- [Result] Sondak VK, King DW, Zager JS, Schneebaum S, Kim J, Leong SP, Faries MB, Averbook BJ, Martinez SR, Puleo CA, Messina JL, Christman L, Wallace AM. Combined analysis of phase III trials evaluating [(9)(9)mTc]tilmanocept and vital blue dye for identification of sentinel lymph nodes in clinically node-negative cutaneous melanoma. Ann Surg Oncol. 2013 Feb;20(2):680-8. doi: 10.1245/s10434-012-2612-z. Epub 2012 Oct 3. PMID 23054107

RESULTS

PARTICIPANT FLOW:
Groups:
- Lymphoseek, Lymphatic Mapping, Injection: Melanoma and breast cancer patients to receive a single dose of 50 µg Lymphoseek radiolabeled with 0.5 or 2.0 mCi Tc 99m and blue dye for lymphatic mapping and surgical resection of lymph nodes.
Period: Overall Study
Arm/Group | Lymphoseek, Lymphatic Mapping, Injection
Started | 163
Completed | 152
Not Completed | 11

BASELINE CHARACTERISTICS:
Population: Of the 163 participants who enrolled in the trial, 153 were administered the study agent, Lymphoseek, and therefore this participant number is used for the baseline analysis.
Groups:
- Lymphoseek: Enrolled patients who were administered any injection of Lymphoseek.
Arm/Group | Lymphoseek
Number analyzed (Participants) | 153
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 101
  >=65 years | 52
Age Continuous [Mean (Standard Deviation); unit: years] | 59.3 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104
  Male | 49
Region of Enrollment [Number; unit: participants]
  United States | 153

OUTCOME MEASURES:

1. Primary Outcome: Concordance of Blue Dye and Lymphoseek
Description: The proportion of lymph nodes detected intraoperatively by blue dye that were also detected by Lymphoseek.
Time Frame: Surgery after injections of Lymphoseek and blue dye
Population: All enrolled patients who were injected with both Lymphoseek and blue dye, who underwent surgery and had at least one lymph node stained intraoperatively by blue dye, and for whom the tissue type (lymphatic/non-lymphatic) and pathology status (presence/absence of tumor cells) was confirmed.
Measure: Number (95% Confidence Interval); unit: Proportion of Lymph Nodes
Units Other Than Participants: Lymph Nodes
Groups:
- Intent-To-Treat: Participants received a single dose of 50 μg Lymphoseek radiolabeled with 0.5 or 2.0 mCi Tc 99m and blue dye for lymphatic mapping and surgical resection of lymph nodes.
Arm/Group | Intent-To-Treat
Number analyzed (Participants) | 133
Number analyzed (Lymph Nodes) | 229
Proportion of Lymph Nodes | 1.0000 [0.9840 to 1.0000]

2. Secondary Outcome: Reverse Concordance of Blue Dye and Lymphoseek
Description: The proportion of lymph nodes detected intraoperatively by Lymphoseek that were also detected by blue dye.
Time Frame: Surgery after injections of Lymphoseek and blue dye
Population: All enrolled patients who were injected with both Lymphoseek and blue dye, who underwent surgery and had at least one lymph node detected by Lymphoseek (at ≥ 3σ count) in vivo, and for whom the tissue type (lymphatic/non-lymphatic) and pathology status (presence/absence of tumor cells) was confirmed.
Measure: Number (95% Confidence Interval); unit: Proportion of Lymph Nodes
Units Other Than Participants: Lymph Nodes
Groups:
- Reverse Intent-To-Treat: Participants received a single dose of 50 μg Lymphoseek radiolabeled with 0.5 or 2.0 mCi Tc 99m and blue dye for lymphatic mapping and surgical resection of lymph nodes.
Arm/Group | Reverse Intent-To-Treat
Number analyzed (Participants) | 152
Number analyzed (Lymph Nodes) | 378
Proportion of Lymph Nodes | 0.6058 [0.5546 to 0.6554]

ADVERSE EVENTS:
Arm/Group | Lymphoseek
Serious Adverse Events (participants affected / at risk) | 8/153
Other Adverse Events (participants affected / at risk) | 0/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lymphoseek (N=153)
Bradycardia (Cardiac disorders) | 1 (1) — Not related to Lymphoseek.
Tachycardia (Cardiac disorders) | 1 (1) — Not related to Lymphoseek.
Cellulitis (Infections and infestations) | 2 (2) — Not related to Lymphoseek.
Herpes Zoster Ophthalmic (Infections and infestations) | 1 (1) — Not related to Lymphoseek.
Seroma (Injury, poisoning and procedural complications) | 1 (1) — Not related to Lymphoseek.
Syncope (Nervous system disorders) | 1 (1) — Not related to Lymphoseek.
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Not related to Lymphoseek.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI shall not submit a publication to journals or professional societies without the prior written approval of the Sponsor.